CLINICAL TRIAL: NCT03116230
Title: Analysis of Pain, Function, and Joint Mechanics in Response to Two Treatments for Knee Pathology
Brief Title: Gait Modification Treatments for Knee Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Peter Andriacchi, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 40688
Record Dates: First submitted 2017-04-11; First posted 2017-04-17 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Knee Injuries; Knee Osteoarthritis
Keywords: Knee pathology
MeSH Terms: conditions — Knee Injuries; Osteoarthritis, Knee | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be told only that we are comparing two types of treatment for their knee pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment A then B (Experimental): Subjects will receive two treatments: (1) a non-invasive external Cutaneous Stimulation device placed on the leg of the subject consisting of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback (vibration) to the subject and (2) a commercially-available knee sleeve, separated by a washout period.
  Interventions: Device: Cutaneous Stimulation; Device: Knee Sleeve
- Experimental Treatment B then A (Experimental): Subjects will receive two treatments: (1) a commercially-available knee sleeve and (2) a non-invasive external Cutaneous Stimulation device placed on the leg of the subject consisting of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback (vibration) to the subject, separated by a washout period.
  Interventions: Device: Cutaneous Stimulation; Device: Knee Sleeve

INTERVENTIONS:
Device: Cutaneous Stimulation — A non-invasive external device that will be placed on the leg of the subject. The device consists of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback to the subject.
Device: Knee Sleeve — Commercially-available knee sleeve.

SUMMARY:
The objective of this study is complete a longitudinal cross-over clinical study to investigate the effect of treatments for knee pathology, including cutaneous stimulation (skin vibration and soft knee brace), on locomotion tasks (i.e. walking, jogging, stair ascending and descending), muscle function, and pain/function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Ambulatory
* Symptomatic knee pain ≥ 3/10 on most of the past 30 days
* Prior ACL injury/surgery, meniscus injury/surgery, and/or physician-diagnosed medial compartment knee osteoarthritis (KL grade 1-3)
* Agreement and ability to use provided interventions during the study period (suggested cumulative wear time during walking of 1-2 hr/day)
* Committed to not starting any new therapies for knee condition during the trial, other than rescue pain medication.

Exclusion Criteria:

* Use of walking aid (e.g. cane, crutch, walker, or wheelchair)
* BMI ≥ 35 kg/m2
* Injection in the affected knee during the previous three months
* Known neuropathy due to diabetes or other causes
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Andriacchi, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Treatment A Then B: Subjects will receive two treatments: (1) a non-invasive external Cutaneous Stimulation device placed on the leg of the subject consisting of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback (vibration) to the subject and (2) a commercially-available knee sleeve, separated by a washout period.
  Cutaneous Stimulation: A non-invasive external device that will be placed on the leg of the subject. The device consists of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback to the subject.
  Knee Sleeve: Commercially-available Passive Knee Bands.
Period: Overall Study
Arm/Group | Experimental Treatment A Then B | Experimental Treatment B Then A
Started | 19 | 19
Completed | 15 | 17
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: All participants entered into the study (all participants received both Treatments A and B in this cross-over study design)
Groups:
- All Participants: Subjects received two treatments assigned in random order: (1) a commercially-available knee sleeve and (2) a non-invasive external Cutaneous Stimulation device placed on the leg of the subject consisting of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback (vibration) to the subject, separated by a washout period.
  Cutaneous Stimulation: A non-invasive external device that will be placed on the leg of the subject. The device consists of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback to the subject.
  Knee Sleeve: Commercially-available knee sleeve.
Arm/Group | All Participants
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38
Peak Knee Flexion Moment (%Bw*Ht) [Mean (Standard Deviation); unit: %Bw*Ht] — The peak knee flexion moment during stance phase of gait, collected during motion capture analysis at a self-selected normal walking speed. The peak knee flexion moment is normalized to percentage body weight and height (%Bw*Ht).
  %Bw*Ht | 3.14 (1.31)
KOOS Pain [Mean (Standard Deviation); unit: units on a scale] — Pain subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
  units on a scale | 66.25 (13.4)
KOOS Symptoms [Mean (Standard Deviation); unit: units on a scale] — Symptom subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
  units on a scale | 59.8 (15.58)
KOOS Function [Mean (Standard Deviation); unit: units on a scale] — Function subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
  units on a scale | 72.31 (15.98)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Knee Flexion Moment (%Bw*Ht)
Description: Within-subject change (follow-up - baseline) in peak knee flexion moment (%Bodyweight*Height) with the intervention at 4-week follow-up versus control (without the intervention) at baseline.
Time Frame: Baseline and 4 week follow-up
Population: Participants completing the study protocol.
Measure: Mean (Standard Deviation); unit: %Bw*Ht
Groups:
- Treatment A (Cutaneous Stimulation): Cutaneous Stimulation: A non-invasive external device that will be placed on the leg of the subject. The device consists of a sensing module to determine specific points in the gait cycle, a processor to analyze signal from the sensor, and a stimulus module to provide feedback to the subject.
- Treatment B (Knee Sleeve): Knee Sleeve: Commercially-available Passive Knee Bands.
Arm/Group | Treatment A (Cutaneous Stimulation) | Treatment B (Knee Sleeve)
Number analyzed (Participants) | 32 | 32
%Bw*Ht | 0.197 (0.374) | 0.018 (0.725)
Statistical Analysis 1: Comparison: Treatment A (Cutaneous Stimulation); Test type: Other; p = 0.005, t-test, 2 sided; Treatment A vs Control
Statistical Analysis 2: Comparison: Treatment B (Knee Sleeve); Test type: Other; p = 0.64, t-test, 2 sided; Treatment B vs Control

2. Secondary Outcome: Change in Pain
Description: Within-subject change (follow-up - baseline) in pain (KOOS sub-scale) with the intervention at 4-weeks versus control (without the intervention) at baseline. KOOS scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Time Frame: Baseline and 4 week follow-up
Population: Participants completing the study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A (Cutaneous Stimulation) | Treatment B (Knee Sleeve)
Number analyzed (Participants) | 32 | 32
units on a scale | 1.476 (12.286) | -0.391 (9.714)

3. Secondary Outcome: Change in Function
Description: Within-subject change (follow-up - baseline) in function (KOOS sub-scale) with the intervention at 4-weeks versus control (without the intervention) at baseline. KOOS scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Time Frame: Baseline and 4 week follow-up
Population: Participants completing the study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A (Cutaneous Stimulation) | Treatment B (Knee Sleeve)
Number analyzed (Participants) | 32 | 32
units on a scale | 4.48 (12.56) | 0.64 (7.903)

4. Secondary Outcome: Change in Symptoms
Description: Within-subject change (follow-up - baseline) in symptoms (KOOS sub-scale) with the intervention at 4-weeks versus control (without the intervention) at baseline. KOOS scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Time Frame: Baseline and 4-week follow-up
Population: Participants completing the study protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A (Cutaneous Stimulation) | Treatment B (Knee Sleeve)
Number analyzed (Participants) | 32 | 32
units on a scale | 3.571 (9.47) | -0.781 (10.876)

ADVERSE EVENTS:
Time Frame: During active study participation, up to 4 weeks for each treatment
Arm/Group | Treatment A (Cutaneous Stimulation) | Treatment B (Knee Sleeve)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 2/32 | 0/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (Cutaneous Stimulation) (N=32) | Treatment B (Knee Sleeve) (N=32)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 0 — Skin irritation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03116230/Prot_SAP_000.pdf